CLINICAL TRIAL: NCT03603041
Title: The Effect of Protein and Omega-3 Fatty Acid Supplementation on Body Composition, Sleep, Cardiometabolic Health and Strength in Postmenopausal Women
Brief Title: Nutrition, Body Composition, and Sleep
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UArkansasFayetteville
Record Dates: First submitted 2018-07-15; First posted 2018-07-27 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Sleep; Body Composition; Strength; Insulin Sensitivity; Energy Expenditure
MeSH Terms: conditions — Insulin Resistance | interventions — Whey Proteins; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): These participants will maintain their daily food and exercise routine and will receive no intervention.
- Whey Protein Supplementation (Experimental): Participants will receive protein supplementation daily for 16 weeks.
  Interventions: Dietary Supplement: Whey protein
- Omega-3 Fatty Acids (O3FA) (Experimental): Participants will receive O3FA supplementation daily for 16 weeks.
  Interventions: Dietary Supplement: Omega-3 fatty acids
- Whey Protein and O3FA (Experimental): Participants will receive protein and O3FA supplementation daily for 16 weeks.
  Interventions: Dietary Supplement: Whey protein; Dietary Supplement: Omega-3 fatty acids
- Whey Protein and Placebo Fat Source (Placebo Comparator): Participants will receive protein and placebo fat source supplementation daily for 16 weeks.
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Participants in the protein arms will receive whey protein daily for 16 weeks.
  Arms: Whey Protein Supplementation; Whey Protein and O3FA; Whey Protein and Placebo Fat Source
Dietary Supplement: Omega-3 fatty acids — Participants in the omega-3 fatty acid arms will receive capsules daily for 16 weeks.
  Arms: Omega-3 Fatty Acids (O3FA); Whey Protein and O3FA

SUMMARY:
The purpose of the research is to determine if protein and omega-3 fatty acid supplementation improve sleep, improve body composition, and improve markers of metabolic health in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

- Postmenopausal women (12+ months following last reported menstrual cycle)

Exclusion Criteria:

* food allergies
* diet restrictions
* do not habitually eat breakfast
* picky eaters\regularly consume protein or omega-3 related supplements
* consume omega-3 fatty acid rich fish (tuna, salmon, etc.) greater than two times per month -have any other diet-related conditions that would prevent them from consuming whey protein supplements and/or omega-3 fatty acid supplements
* smoking
* habitual alcohol consumption (> 4 drinks/week)
* medication impacting appetite or metabolism
* Lipid or blood pressure lowering medication
* Hormone replacement therapy

Max Age: 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | Change in sleep quality from baseline (day 0) to 16 weeks.
  Pittsburgh Sleep Quality Index (PSQI) will assess sleep quality and disturbance. This is a elf-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

SECONDARY OUTCOMES:
Dietary intake | Change in dietary intake from baseline (day 0) to 16 weeks.
  Dietary intake will be measured using 3-day, weighed food records.
Sleep Quantity | Change in sleep quantity from baseline (day 0) to 16 weeks.
  Sleep duration will be measured using Actigraph monitors worn on the wrist.
Body composition | On day 1 and day 112 (final day of 16-week intervention) of study.
  Body composition will be measured using dual x-ray absorptiometry (DEXA).
Resting energy expenditure (REE) | On day 1 and day 112 (final day of 16-week intervention) of study.
  REE will be measured using indirect calorimetry.
Orexin | On day 1 and day 112 (final day of 16-week intervention) of study.
  Intravenous blood samples will be collected and orexin measured using a commercial kit.

OTHER OUTCOMES:
Mood | Change in sleep quality from baseline (day 0) to 16 weeks.
  Mood will be assessed using the Profile of Mood States (POMS) questionnaire. The POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A five-point scale ranging from "not at all" to "extremely" is used to assess participant mood states.
Strength | On day 1 and day 112 (final day of 16-week intervention) of study.
  Strength will be assessed using a standard hand-grip dynamometer .
Glucose | On day 1 and day 112 (final day of 16-week intervention) of study.
  Intravenous blood samples will be collected and glucose measured using a commercial kit.
Insulin | On day 1 and day 112 (final day of 16-week intervention) of study.
  Intravenous blood samples will be collected and insulin measured using a commercial kit.
Blood lipids | On day 1 and day 112 (final day of 16-week intervention) of study.
  Intravenous blood samples will be collected and blood lipids measured using a commercial kit.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie I Baum, Phd, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No